CLINICAL TRIAL: NCT00595478
Title: Family Based Contingency Management for Adolescent Alcohol Abuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Catherine Stanger, Associate Professor, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 85846; 1R01AA016917-01 (NIH); 1R01AA016917-02 (NIH); 1R01AA016917-03 (NIH)
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Results first posted 2018-03-29 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Alcohol Abuse
MeSH Terms: conditions — Alcoholism | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Motivational Enhancement Therapy (MET)/CBT+CM/BPT
  Interventions: Behavioral: Motivational Enhancement Therapy (MET)/CBT+CM
- 2 (Active Comparator): Motivational Enhancement Therapy (MET)/CBT
  Interventions: Behavioral: Motivational Enhancement Therapy (MET)/CBT

INTERVENTIONS:
Behavioral: Motivational Enhancement Therapy (MET)/CBT+CM — Behavioral Treatment
  Arms: 1
Behavioral: Motivational Enhancement Therapy (MET)/CBT — Behavioral Treatment
  Arms: 2

SUMMARY:
The goal is to adapt the family-based CM treatment to target primary adolescent alcohol abuse and dependence.

Specific Aim 1 is to provide a preliminary demonstration of the efficacy of a family-based CM intervention to treat adolescent alcohol abuse and dependence. CM components include:

1. an incentive program to enhance the adolescent's engagement in the treatment process and engender alcohol abstinence by providing positive reinforcement for documented abstinence via breathalyzers administered by parents regularly at home, self and parent report, and clinic-based urine drug testing; and
2. a parent management training program to enhance and maintain the positive effects of the incentive program by teaching parents how to effectively use contingency management in the home environment to motivate their adolescent to achieve abstinence and improve their behavior in other domains.

A randomized trial will determine whether the CM intervention enhances outcomes when added to a standard individual cognitive behavioral therapy (CBT).

Specific Aim 2 is to determine whether and how treatment interventions modify parental and adolescent risk and protective factors using observational and laboratory measures (parenting practices, family functioning, risk taking, delay discounting, and child and parent psychopathology) and to determine whether these factors are associated with outcomes over time.

Specific Aim 3 is to test gene x environment (treatment) interactions in adolescent substance abuse. Findings will extend the scientific evidence for CM and support the ability of parents to implement CM at home. Findings that support the CM model's efficacy will make a significant contribution to research on the treatment of adolescent alcohol abuse, which has lagged behind research on adult substance abuse and on adolescent illicit drug use.

DETAILED DESCRIPTION:
Approximately 1.5 million youth ages 12-17 (representing 6.1% of all youth in that age range) are in need of treatment for alcohol abuse, yet only 7.2% of those in need of treatment received it. Importantly, most youth (90.5%) who were classified as needing treatment based on their self report of Adolescent Alcohol Study Plan; v.2; 3/30/12Page 2 of 35 symptoms, perceived no need for treatment. Thus, there is a need to develop treatments that target populations of alcohol abusing youth who are not highly motivated to change their substance use. New outpatient family based and contingency management interventions for adolescent marijuana abuse have been developed, yet none of these interventions has specifically targeted adolescent alcohol use. It is important to target primary alcohol abuse and dependence in adolescence as approximately 20% of treatment-seeking youth report primary problems with alcohol. The primary aim of this proposal is to adapt our family-based contingency-management treatment to target adolescent alcohol abuse and dependence. This project will develop, manualize, and pilot a contingency management intervention that includes two components. First, an incentive program will enhance the adolescent's engagement in the treatment process and engender alcohol abstinence by providing positive reinforcement for documented abstinence via breathalyzers administered by parents regularly at home, self and parent report, and clinic based urine drug testing. Second, a parent management training program will enhance and maintain the positive effects of the incentive program by teaching parents how to effectively use contingency management in the home environment to motivate their adolescent to achieve abstinence and improve their behavior in other domains.

ELIGIBILITY:
Inclusion Criteria:

* 12-18 years old (if 18, must attend high school and live at home)
* Report using alcohol during the previous 30 days
* Have a parent/guardian who can participate
* Meet DSM criteria for either Alcohol Abuse or Dependence
* Youth who meet DSM criteria for Alcohol Dependence may also meet criteria for Marijuana Abuse or Dependence and other Drug Abuse
* Youth who meet DSM criteria for Alcohol Abuse, may also meet criteria for Marijuana or other Drug Abuse
* Live within a 30-minute drive of the clinic

Exclusion Criteria:

* Meet DSM criteria for Drug Dependence (other than Marijuana Dependence)
* Meet DSM criteria for Alcohol Abuse with Marijuana Dependence. Use of other drugs will not be excluded
* Participants will also be excluded if they exhibit an active psychosis
* Have a severe medical or psychiatric illness that will limit participation
* Are pregnant or breast-feeding

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 75 (Actual)
Dates: Start 2007-08; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Stanger, Ph.D., Principal Investigator — Dartmouth College
Locations (1):
- Geisel School of Medicine at Dartmouth, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stanger C, Scherer EA, Babbin SF, Ryan SR, Budney AJ. Abstinence based incentives plus parent training for adolescent alcohol and other substance misuse. Psychol Addict Behav. 2017 Jun;31(4):385-392. doi: 10.1037/adb0000279. Epub 2017 Apr 17. PMID 28414474

RESULTS

PARTICIPANT FLOW:
Groups:
- (MET)/CBT+CM/BPT: Motivational Enhancement Therapy (MET)/CBT+CM/BPT
  Motivational Enhancement Therapy (MET)/CBT+CM: Behavioral Treatment
- (MET)/CBT: Motivational Enhancement Therapy (MET)/CBT
  Motivational Enhancement Therapy (MET)/CBT: Behavioral Treatment
Period: Treatment
Arm/Group | (MET)/CBT+CM/BPT | (MET)/CBT
Started | 37 | 38
Completed | 37 | 38
Not Completed | 0 | 0
Period: 36-week Follow-up Period
Arm/Group | (MET)/CBT+CM/BPT | (MET)/CBT
Started | 37 | 38
Completed | 28 | 30
Not Completed | 9 | 8
Not completed — Lost to Follow-up | 5 | 4
Not completed — Withdrawal by Subject | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | (MET)/CBT+CM/BPT | (MET)/CBT | Total
Number analyzed (Participants) | 37 | 38 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.1 (1.2) | 16.2 (1.2) | 16.1 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 27 | 29 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 29 | 32 | 61
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37 | 38 | 75
Tobacco user [Count of Participants; unit: Participants] | 30 | 30 | 60
Mean intake proportion of days used alcohol in past 30 days [Mean (Standard Deviation); unit: proportion of days used alcohol] — We report the proportion of days used because not all participants provided data for the identical number of days at each assessment. Therefore the denominator differs across participants, and the proportion of days on which use was reported is the more appropriate measure of use frequency.
  proportion of days used alcohol | 0.12 (0.16) | 0.12 (0.14) | 0.12 (0.15)
Mean drinks per drinking day [Mean (Standard Deviation); unit: Drinks] | 5.7 (4.9) | 6.4 (4.5) | 6.0 (4.7)
DSM Alcohol Use Disorder [Count of Participants; unit: Participants]
  Dependence | 7 | 7 | 14
  Abuse only | 12 | 14 | 26
  None | 18 | 17 | 35

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Abstinence
Description: Number of non-abstinent urinalysis (ETG-positive) samples during 14 weeks of treatment (considering missing samples as non-abstinent)
Time Frame: Weekly up to 14 weeks
Measure: Mean (Standard Deviation); unit: Samples
Arm/Group | (MET)/CBT+CM/BPT | (MET)/CBT
Number analyzed (Participants) | 37 | 38
Samples | 2.9 (3.5) | 2.6 (3.6)
Statistical Analysis 1: Comparison: (MET)/CBT+CM/BPT vs (MET)/CBT; Test type: Superiority; p = 0.66, Poisson regression; Chi-square test with 1 degree of freedom; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.29 to 2.18] — Odds ratio for 0 ETG-positive samples for MET/CBT+CM/BPT (numerator) vs. MET/CTB (denominator)
Statistical Analysis 2: Comparison: (MET)/CBT+CM/BPT vs (MET)/CBT; Test type: Superiority; p = 0.61, Poisson regression; Chi-square test with 1 degree of freedom; mean ratio = 0.93, 95% CI 2-sided [0.71 to 1.22] — Mean ratio for number of ETG-positive samples, if >0 ETG-positive samples: MET/CBT+CM/BPT (numerator) vs. MET/CTB (denominator)

2. Secondary Outcome: Days of Alcohol Use During 36-week Follow-up Period
Description: Percentage of days alcohol used during the 36-week follow-up period after treatment ended measured via timeline follow-back.
Time Frame: Monthly up to 9 months (36 weeks)
Population: The analysis population consisted of only participants with follow-up (alcohol use) data on at least 85% of the days in the 36-week follow-up period.
Measure: Mean (Standard Deviation); unit: percentage of days used
Arm/Group | (MET)/CBT+CM/BPT | (MET)/CBT
Number analyzed (Participants) | 28 | 30
percentage of days used | 5.6 (8.8) | 7.6 (10.6)
Statistical Analysis 1: Comparison: (MET)/CBT+CM/BPT vs (MET)/CBT; Test type: Superiority; p = 0.74, Poisson regression; Chi-square test with 1 degree of freedom; Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.26 to 2.62] — Odds ratio for 0% days using alcohol during the 36 week follow-up period: MET/CBT+CM/BPT (numerator) vs. MET/CTB (denominator)
Statistical Analysis 2: Comparison: (MET)/CBT+CM/BPT vs (MET)/CBT; Test type: Superiority; p = 0.007, Poisson regression; Chi-square test with 1 degree of freedom; mean ratio = 0.74, 95% CI 2-sided [.59 to .92] — Mean ratio for percentage of days with alcohol use during the 36 week follow-up period, if alcohol was used: MET/CBT+CM/BPT (numerator) vs. MET/CTB (denominator)

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | (MET)/CBT+CM/BPT | (MET)/CBT
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/38
Other Adverse Events (participants affected / at risk) | 0/37 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No